CLINICAL TRIAL: NCT04151498
Title: Project RAMP (Reengagement and Assessment Mobile Program): A Field Visit Model for HIV Clinic Reengagement
Brief Title: HIV Reengagement and Assessment Mobile Program (Project RAMP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-0664
Record Dates: First submitted 2019-10-23; First posted 2019-11-05 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): This group will complete an HIV health reengagement intervention on a mobile van, in addition to a pre- and post-intervention qualitative interview.
  Interventions: Behavioral: Reengagement and Assessment Mobile Program; Other: Qualitative Interview
- Usual Care Reengagement Group (Other): This group will complete a qualitative interview about barriers and facilitators to HIV care.
  Interventions: Other: Qualitative Interview
- Non-enrolling Group (No Intervention): This group will not be enrolled in the intervention, and will include de-identified data from clinic patients referred to bridge counselors during the study time period that do not participate in the intervention.

INTERVENTIONS:
Behavioral: Reengagement and Assessment Mobile Program — Participants will participate in mobile clinic visit that will include an educational interview, adherence counseling, and standard blood draws for HIV reengagement. The goal of this intervention is to motivate participants to become reengaged in traditional HIV care by making an in person clinic appointment.
  Other Names: Project RAMP
  Arms: Intervention Group
Other: Qualitative Interview — Qualitative interview about barriers and facilitators to HIV care, and experience at most recent clinic visit.
  Arms: Intervention Group; Usual Care Reengagement Group

SUMMARY:
The North Carolina Bridge Counselor system is designed to help link out of care HIV positive patients back into HIV care. It has improved initial linkages and patient re-engagement overall, but for a sizable group of patients, the current system has not been effective, leaving a population of hard-to-reach, lost-to-care patients who remain out of care. There is limited understanding of the lived experiences of patients who fall out of HIV care and become recalcitrant to re-engagement because they are difficult to reach and therefore underrepresented in research. Out of care HIV+ patients who have not reengaged in care following the standard of care who chose to enroll in the study will participate in 2 semi-structured interviews and receive a field-based HIV re-engagement and treatment intervention (Project RAMP). Project RAMP will consist of up to 4 visits from an outreach research nurse designed to serve as an "on-ramp" to HIV care. At these visits, the outreach number will counsel on HIV care and treatment and obtain a medical history and labs. Results will be communicated to the participant's clinic provider in an effort to both encourage the patient to return to care and facilitate more rapid antiretroviral therapy (ART) initiation by the clinic provider. The research team will also provide the participant in-person assistance with scheduling a clinic visit. Clinic providers may re-initiate ART prior to the reengagement clinic visit, with adherence support provided by the outreach nurse.

DETAILED DESCRIPTION:
The overall purpose of the Project RAMP intervention is to find out what challenges make it hard for people living with HIV to keep their in-person clinic appointments. The investigators also hope to learn how much a mobile HIV treatment van may help patients who have been out of care for a minimum of 6 months, to re-start keeping regular clinic visits. The investigators also hope this information will help be useful in learning best practices for providing health care to people living with HIV.

This study will recruit a total of 30 participants, 20 for the intervention and 10 for the usual care group. Participants will be recruited through bridge counselors at the partnering clinic, whose roles and responsibilities consist of finding and reaching out to patients who have been out of HIV care in an attempt to get them reengaged.

Participants will have up to 5 study visits that are between 1- 4 weeks apart. Each visit will last about 1 to 1.5 hours. Participants will also be asked to participate in two in depth interview: a baseline interview at the start of the study that will ask questions about each participant's experience with their past clinic visits and an exit interview at the end of the study regarding their experience participating in the HIV mobile treatment program (Project RAMP). The pre-intervention visit (Visit 0) includes the first interview, providing some brief information about you, a urine pregnancy test for participants who are female, and a brief meeting with a financial technician who will help participants complete their insurance information. Intervention Visit 1 will include a nurse from the partnering clinic administering the video educational intervention, HIV medication adherence counseling, a health history form, blood draws for standard reengagement labs (CD4 count, HIV viral load, comprehensive metabolic panel, complete blood count with differential, rapid plasma reagin and HIV genotype). Specimens from these visits will be delivered to partnering clinic for analysis. Notes from the mobile visit will be shared with the study PI, who will in term communicate these notes with the assigned clinic provider of each participant. Visits 2-4 will include a study nurse conducting additional blood draws if recommended by their assigned provider, and a review of adherence counseling and health history forms.

At the end of each intervention visit, participants will be if they would like to make an in person clinic appointment. Those who decline at the end of intervention Visits 1-3 will be offered an additional field visit appointment. Those who decline an in person clinic appointment at the end of Visit 4 will move on to completing the exit interview in person at this time and will complete the study following the exit interview. Participants who schedule a clinic appointment will have their exit interview in person or via phone within 3 months of their clinic visit. All participants will be follow up to 6 months after their last study visit to to access their viral load, if this information is available.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* HIV positive
* Referred to the bridge counselors by the partnering clinic as out of care for >=6 months and not successfully re-engaged in care by a bridge counselor
* Willing and able to give informed consent and adhere to study visits

Exclusion Criteria:

* Unwilling or physically unable to participate in study visits on the mobile van
* Lack of English language fluency
* Planning or preferring to transfer HIV care to an HIV clinic other than the partnering HIV clinic
* Pregnant women will be expedited into clinical care and will not be eligible for the study
* Presence of mobility or balance issues that prevent patient from safely stepping up onto the mobile unit without assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible persons screened that enroll. | Screening call through Visit 0 when consent occurs, approximately 2 - 3 weeks
  Percentage of all eligible persons that are screened by the study team that enroll in Project RAMP during the intervention period.
Qualitative Summary of Participants' Experiences from In-depth Baseline Interview | Up to approximately 1 hour at Baseline
  Data will be obtained from in-depth qualitative interviews. Summary will include reasons why patients who have been out of care for more than 6 months have been lost to care.
Qualitative Summary of Participants' Experiences from In-depth Exit Interview | Up to approximately 1 hour at Exit Interview
  Data will be obtained from in-depth qualitative interviews. Summary will include information evaluating participants' experiences in Project RAMP.

SECONDARY OUTCOMES:
Number of participants who are successfully reengaged following the intervention. | 6 months following the participants' last intervention visit
  Reengagement is defined as 1 kept visit following the intervention. The investigators will collect this data from the participants' medical record.
Number of participants who are successfully retained following the intervention. | 6 months following the participants' last intervention visit
  Retention is defined as 2 kept visits following the intervention. The investigators will collect this data from the participant's medical record.
Number of participants who have viral suppression following the intervention. | 6 months following participants' last intervention visit
  Viral suppression is defined as <200 copies/mL. The investigators will collect data on viral suppression from participant's medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sellers, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 9 to 36 months following publication.
Access Criteria: Deidentified individual data that supports the results will be shared provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.